CLINICAL TRIAL: NCT05002296
Title: Effect of Rotatory Upper Cervical Manipulation on Reflex Cervical Vertigo in Chronic Mechanical Neck Pain Patients
Brief Title: Effect of Rotatory Upper Cervical Manipulation on Reflex Cervical Vertigo
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Ramy Salama Draz, lecturer of physiotherapy, cairo university, Cairo University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P.T.REC/012/002663
Record Dates: First submitted 2021-06-26; First posted 2021-08-12 (Actual); Last update posted 2021-08-12 (Actual); Status verified 2021-08

CONDITIONS: Vertigo
MeSH Terms: conditions — Vertigo

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- traditional physical therapy program (Active Comparator)
  Interventions: Procedure: upper cervical manipulation
- rotatory upper cervical manipulation to both sides (Experimental)
  Interventions: Procedure: upper cervical manipulation

INTERVENTIONS:
Procedure: upper cervical manipulation — rotatory upper cervical manipulation to both sides. The treatment program was conducted for twelve sessions (three sessions per week). Assessment procedures were performed before and after treatment through visual analogue scale (VAS)

SUMMARY:
Cervical reflex vertigo is a non-common cause of vertigo, caused by decreased afferent input from the upper three cervical segments to vestibular nuclei.

ELIGIBILITY:
Inclusion Criteria:

* cervical pain
* vertigo

Exclusion Criteria:

* severe osteoporosis
* blood circulation problem

Max Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 40 (Estimated)
Dates: Start 2021-06-15 (Actual); Primary Completion 2021-09 (Estimated); Study Completion 2021-10 (Estimated)

PRIMARY OUTCOMES:
pain intensity seems to be improved | 3 monthes
  Assessment procedures were performed before and after treatment through visual analogue scale (VAS)
vertigo seems to be significantly improved | 3 monthes
  Dix-Hallpike test was used to asses the vertigo degree and improvement within and after the treatment programme

CONTACTS AND LOCATIONS:
Overall Officials: Abdelaziz Elsherif, lecturer, Study Director — lecturer at faculty of physiotherapy, Cairo university; Amr Hassan, professor, Study Director — professor at faculty of medicine
Locations (1):
- faculty of physical therapy Cairo university, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided